CLINICAL TRIAL: NCT00975182
Title: A Phase Ib, Open-Label, Dose-Escalation Study of the Safety and Pharmacology of GDC-0941 in Combination With Erlotinib in Patients With Advanced Solid Tumors
Brief Title: A Study of the Safety and Pharmacology of GDC-0941 in Combination With Erlotinib in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GDC4626g; GO01301 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2009-09-08; First posted 2009-09-11 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer, Solid Cancers
Keywords: PI3K; NSCLC; Tarceva
MeSH Terms: interventions — 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine; Erlotinib Hydrochloride

ARMS (1):
- A (Experimental)
  Interventions: Drug: GDC-0941; Drug: erlotinib HCl

INTERVENTIONS:
Drug: GDC-0941 — Oral repeating dose
Drug: erlotinib HCl — Oral repeating dose

SUMMARY:
This is an open-label, multicenter, Phase Ib dose-escalation study to assess the safety, tolerability, and pharmacokinetics (PK) of oral (PO) GDC-0941 administered in combination with PO erlotinib in patients with advanced solid tumors and patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) who have failed at least one prior chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Documented locally advanced or metastatic solid tumors for which standard therapy either does not exist or has proven ineffective or intolerable (dose-escalation stage only)
* Documented locally advanced or metastatic NSCLC in patients who have failed at least one prior chemotherapy-based regimen for incurable disease (cohort-expansion stage only)
* Adequate organ function as assessed by laboratory tests
* Evaluable disease or disease measurable per Response Evaluation Criteria in Solid Tumors (RECIST)
* Agreement to use an effective form of contraception for the duration of the study

Exclusion Criteria:

* Any anti-cancer therapy (e.g., chemotherapy, biologic therapy, or hormonal therapy) within a specified timeframe prior to first study treatment
* Prior treatment with PI3K pathway-inhibiting agents (cohort-expansion stage only)
* History of Grade >= 3 fasting hyperglycemia or diabetes requiring regular medication
* Current clinically significant and uncontrolled systemic disease (e.g., cardiovascular, pulmonary, or metabolic)
* History of clinically significant cardiac or pulmonary dysfunction
* History of malabsorption syndrome or other condition that would interfere with enteral absorption
* Clinically significant history of liver disease
* Any condition requiring full-dose anticoagulants, such as warfarin, heparin, or thrombolytic agents
* Active autoimmune disease and/or need for corticosteroid therapy
* Known brain metastases that are untreated, symptomatic, or require therapy
* Pregnancy, lactation, or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Incidence, nature, and severity of adverse events | Through study completion or early study discontinuation
Tumor response | Assessed at periodic intervals

SECONDARY OUTCOMES:
PK parameters of GDC-0941 (total exposure, and maximum and minimum serum concentrations) | Through study completion or early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (4):
- United States (2):
  - Aurora, Colorado
  - New Brunswick, New Jersey
- Netherlands (2):
  - Amsterdam
  - Utrecht